CLINICAL TRIAL: NCT01377623
Title: Pilot Study on the Effect of Dexmedetomidine on Inflammatory Responses in Patients Undergoing Lumbar Spinal Fusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10-02185
Record Dates: First submitted 2011-01-03; First posted 2011-06-21 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Spinal Stenosis; Inflammation
Keywords: Spinal fusion; Inflammatory response; Inflammatory markers; Dexmedetomidine
MeSH Terms: conditions — Spinal Stenosis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): Eligible subjects will be randomized to one of the two treatment group in1:1 ratio to receive either DEX or matching placebo (PBO, LR).
  Interventions: Drug: Placebo group
- Dexmedetomidine group (Experimental): Eligible subjects will be randomized to one of the two treatment group in1:1 ratio to receive either DEX or matching placebo (PBO, LR).
  Interventions: Drug: Dexmedetomidine group

INTERVENTIONS:
Drug: Dexmedetomidine group — Subjects undergoing one or two level spinal fusion surgery will be screened for eligibility to participate in the study. Subject will be screened, recruited and randomized during the preadmission visit or the day of surgery. Eligible subjects will be randomized to one of the two treatment group in1:1 ratio to receive either DEX or matching placebo (PBO, LR).
  Arms: Dexmedetomidine group
Drug: Placebo group — Fifty six subjects (28 in each arm) will be enrolled. Subjects undergoing one or two level spinal fusion surgery will be screened for eligibility to participate in the study. Subject will be screened, recruited and randomized during the preadmission visit or the day of surgery. Eligible subjects will be randomized to one of the two treatment group in1:1 ratio to receive either DEX or matching placebo (PBO, LR).
  Arms: Placebo group

SUMMARY:
The aim of the proposed study is to examine the effect of DEX on the inflammatory response in major surgery. More importantly, the investigators will correlate changes in the concentration of inflammatory mediators with meaningful clinical outcomes.

DETAILED DESCRIPTION:
Surgical injury to tissue causes a variety of profound physiologic reactions which are essential for the restoration of an organisms' homeostasis. The inflammatory response involves a surge of stress hormones (i.e. ACTH, cortisol, catecholamines), activation of the complement system, migration of leukocytes to the site of injury, the release of cytokines (i.e. interleukins, tumor necrosis factor), as well as other cellular products (i.e. superoxide radicals, proteases, growth factors) (1-3). An appropriate inflammatory cascade is essential for tissue reconstitution and infection control. The associated impairment of multiple organ function is generally mild, because of the physiological reserve of the biological systems. However, a systemic inflammatory response may also lead to postoperative complications in the elderly, neonates, and patients with significant co-morbidity (4, 5). Indeed, mediators of inflammation may induce fatigue and prolong convalescence in healthy patients. On the other hand, dysregulation or suppression of the inflammatory process may lead to improper wound healing, infection and, as demonstrated recently, even an increase in cancer recurrence due to reduction in natural killer cell activity (6, 7).

Anesthetic management may affect both immunostimulatory and immunosuppressive mechanisms either directly by modulating functions of immune cells or indirectly by attenuating the stress response. For example, inhalational anesthetics inhibit neutrophil function and depress lymphocyte proliferation while increasing pro-inflammatory cytokine levels (8, 9)). Propofol also inhibits neutrophil and monocyte function, and has strong anti-inflammatory and anti-oxidative effects (10). Opioids attenuate the direct cell immune response, but have only minimal effects on systemic inflammatory responses (11). It is expected that the choice of anesthetic technique may disturb the balance between pro- and anti-inflammatory responses thus affecting clinical outcomes. A most advantageous anesthetic choice would enhance or have a neutral effect on cellular immunity while minimizing contribution to the systemic inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (> 18) male or female who will undergo surgery for spinal fusion with general anesthesia.
2. If female, subject is non-lactating and is either:

   * Not of childbearing potential
   * Of childbearing potential but is not pregnant at time of baseline as determined by pre-surgical pregnancy testing.
3. Subject is ASA physical status 1, 2, or 3.

Exclusion Criteria:

1. Cognitively impaired (by history)
2. Subject requires chronic antipsychotic history
3. Subject is anticipated to require an additional surgery within 90 days after the intended spinal fusion
4. Subject known to be in liver failure
5. Subject has received treatment with alpha-2-agonist or antagonist within 2 weeks of study entry
6. Subject for whom opiates, benzodiazepines, DEX are contraindicated
7. Chronic use of steroids/NSAIDs
8. Patients with serious bradycardia related arrhythmias, i.e. 2nd degree block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Bekker, MD, PhD, Principal Investigator — NYU School of Medicine; Michael Urban, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (2):
- United States (2):
  - NYU Langone Medical Center, Department of Anesthesiology, New York, New York
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Bekker A, Haile M, Kline R, Didehvar S, Babu R, Martiniuk F, Urban M. The effect of intraoperative infusion of dexmedetomidine on the quality of recovery after major spinal surgery. J Neurosurg Anesthesiol. 2013 Jan;25(1):16-24. doi: 10.1097/ANA.0b013e31826318af. PMID 22824921

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine Group (PFD): Anesthesia maintained with propofol/fentanyl/dexmedetomidine
- Placebo Group (PFS): Anesthesia maintained with propofol/fentanyl/saline
Period: Overall Study
Arm/Group | Dexmedetomidine Group (PFD) | Placebo Group (PFS)
Started | 33 | 33
Completed | 26 | 28
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Population: Baseline data is only available for those participants who completed the study
Groups:
- Placebo Group: Subjects undergoing one or two level spinal fusion surgery will be screened for eligibility to participate in the study. Subject will be screened, recruited and randomized during the preadmission visit or the day of surgery. Eligible subjects will be randomized to one of the two treatment group in1:1 ratio to receive either DEX or matching placebo (PBO, LR).
- Dexmedetomidine Group: Fifty six subjects (28 in each arm) will be enrolled. Subjects undergoing one or two level spinal fusion surgery will be screened for eligibility to participate in the study. Subject will be screened, recruited and randomized during the preadmission visit or the day of surgery. Eligible subjects will be randomized to one of the two treatment group in1:1 ratio to receive either DEX or matching placebo (PBO, LR).
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Dexmedetomidine Group | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.1) | 55.3 (12.3) | 56.18 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 15 | 21 | 36

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery Score (QoR-40)
Description: The QoR-40 is a 40 item questionnaire in which each question is answered with a score of 1-5. QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Time Frame: Post-operative Day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine Group (PFD) | Placebo Group (PFS)
Number analyzed (Participants) | 26 | 28
units on a scale | 183.04 (2.76) | 169.3 (3.87)

2. Secondary Outcome: Concentration of TNF-alpha
Time Frame: Post-operative Day 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Dexmedetomidine Group (PFD) | Placebo Group (PFS)
Number analyzed (Participants) | 26 | 28
pg/ml | 10.1 [3.8 to 12.7] | 7.9 [2.1 to 11.4]

3. Secondary Outcome: Concentration of IL-1a
Time Frame: Post-operative Day 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Dexmedetomidine Group (PFD) | Placebo Group (PFS)
Number analyzed (Participants) | 26 | 28
pg/ml | 2.52 [1.4 to 3.6] | 2.58 [1.4 to 2.6]

4. Secondary Outcome: Concentration of IL-6
Time Frame: Post-operative Day 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Dexmedetomidine Group (PFD) | Placebo Group (PFS)
Number analyzed (Participants) | 26 | 28
pg/ml | 60.8 [27.3 to 122.8] | 50.0 [11.2 to 82.1]

5. Secondary Outcome: Concentration of IL-8
Time Frame: Post-operative Day 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Dexmedetomidine Group (PFD) | Placebo Group (PFS)
Number analyzed (Participants) | 26 | 28
pg/ml | 20.9 [12.6 to 31.2] | 16.4 [6.2 to 24.6]

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine Group (PFD) | Placebo Group (PFS)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 0/26 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes